CLINICAL TRIAL: NCT06516484
Title: Ropustin for Refractory Aplastic Anaemia After Radiotherapy - a Single-centre, Prospective, Open-label, Single-arm Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LRA-2024-001
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Aplastic Anemia
Keywords: After radiotherapy and chemotherapy; Romiplostim
MeSH Terms: conditions — Anemia, Aplastic | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Romiplostim group (Experimental): Enrolled patients were given roprostin (20 µg/kg subcutaneously once weekly) for at least 3 months, with discontinuation of roprostin for platelet counts ≥50 x 10^9/L and continuation of roprostin for platelet counts <50 x 10^9/L. Responders were continued to 6 months. Responders continue to use the drug until 6 months.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — Enrolled patients were given roprostin (20 µg/kg subcutaneously once weekly) for at least 3 months, with discontinuation of roprostin for platelet counts ≥50 x 10^9/L and continuation of roprostin for platelet counts <50 x 10^9/L. Responders were continued to 6 months. Responders continue to use the drug until 6 months.

SUMMARY:
To investigate the efficacy and safety of roprostin in the treatment of refractory AA after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, male or female.
2. Diagnosis consistent with refractory AA after radiotherapy. refractory is defined as patients who have failed to respond to at least an adequate amount of supportive therapy, cyclosporine or povidone TPO-RA for 3 months .
3. At least one of the following conditions was met at enrolment: haemoglobin <90 g/L. Platelets <30 x 10^9/L, neutrophils <1.0 x 10^9/L.
4. Baseline liver and renal function is less than two times the normal value.
5. No active infection.
6. Agreed to sign the consent form.
7. Eastern Cooperative Oncology Group (ECOG) score of 0-2.

Exclusion Criteria:

1. Other causes of whole blood cytopenia, such as myelodysplastic syndromes (MDS).
2. Presence of cytogenetic evidence of clonal haematological bone marrow disorders (MDS, AML).
3. PNH clones ≥50%.
4. Hematopoietic stem cell transplantation (HSCT) prior to enrolment.
5. Prior treatment with ATG.
6. Infection or bleeding uncontrolled by standard therapy.
7. Allergy to roprostin.
8. Active HIV, HCV or HBV infection or cirrhosis or portal hypertension.
9. Any concomitant malignancy, localised basal cell carcinoma of the skin within 5 years.
10. Previous history of thromboembolic events, heart attack or stroke (including antiphospholipid antibody syndrome) and current use of anticoagulants.
11. Pregnant or lactating (breastfeeding) women.
12. Participation in another clinical trial within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 months, 6 months
  Overall response rate (ORR) is defined as the ratio of complete response (CR) + partial response (PR).CR is defined as a haemoglobin level ≥120 g/L, neutrophil count >1.5 × 10^9/L and platelet count >150 × 10^9/L in patients not receiving transfusion.PR is defined as not transfusion dependent (if previously dependent), or at least one cell lineage doubled or normalised or increased at baseline, or initial ANC < 0.5 x 10^9/L increased by at least 0.5 x 10^9/L after treatment, or initial PLT < 20 x 10^9/L increased by at least 20 x 10^9/L after treatment.
CRR | 3 months, 6months
  Overall response rate (ORR) is defined as the ratio of complete response (CR) + partial response (PR).CR is defined as a haemoglobin level ≥120 g/L, neutrophil count >1.5 × 10^9/L and platelet count >150 × 10^9/L in patients not receiving transfusion.PR is defined as not transfusion dependent (if previously dependent), or at least one cell lineage doubled or normalised or increased at baseline, or initial ANC < 0.5 x 10^9/L increased by at least 0.5 x 10^9/L after treatment, or initial PLT < 20 x 10^9/L increased by at least 20 x 10^9/L after treatment.

SECONDARY OUTCOMES:
safety events | 3 months，6months
  Proportion and severity of adverse events in patients during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Bing Han, PhD, Principal Investigator — Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuter DJ. The biology of thrombopoietin and thrombopoietin receptor agonists. Int J Hematol. 2013 Jul;98(1):10-23. doi: 10.1007/s12185-013-1382-0. Epub 2013 Jul 3. PMID 23821332
- [Background] Lee JW, Lee SE, Jung CW, Park S, Keta H, Park SK, Kim JA, Oh IH, Jang JH. Romiplostim in patients with refractory aplastic anaemia previously treated with immunosuppressive therapy: a dose-finding and long-term treatment phase 2 trial. Lancet Haematol. 2019 Nov;6(11):e562-e572. doi: 10.1016/S2352-3026(19)30153-X. Epub 2019 Aug 29. PMID 31474546